CLINICAL TRIAL: NCT06820450
Title: STERONLINE: Steroidome and Exposome of Endometriosis Single-center Case-control Study
Brief Title: Pilot Study to Characterize the Endometriosis Steroidome and Its Link to Endocrine Disruptors and Vaginal Dysbiosis
Acronym: STERONLINE
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0498
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis
Keywords: Steroidome; exposome; LC-HRMS
MeSH Terms: conditions — Endometriosis | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 10 ml blood sample (2 x 5 ml tubes) and a 20 ml urine sample for steroid profile analysis; A vaginal swab to characterise your microbiota.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1. Controls (n=45): * Women with no laparoscopically confirmed signs of deep endometriosis.
  * No clinico-biological criteria in favour of a diagnosis of endometriotic disease, nor any radiological signs (ultrasound or MRI) suggestive of endometriosis.
  A blood test (2 x 5 ml dry tubes) and a 20 ml urine sample will be taken to analyze steroid profiles, as well as a vaginal sample to characterize the microbiota.
  Interventions: Other: Blood test; Other: urine sample; Other: vaginal sample
- Group 2. Deep endometriosis (n = 90): * 45 patients with endometriome
  * 45 patients without endometriome Deep endometriosis confirmed by surgery or MRI Newly diagnosed women (less than 12 months).
  * Severe, deep-seated endometriotic pathology with surgical indication (clinical examination, imaging tests, pre-operative findings).
  A blood test (2 x 5 ml dry tubes) and a 20 ml urine sample will be taken to analyze steroid profiles, as well as a vaginal sample to characterize the microbiota.
  Interventions: Other: Blood test; Other: urine sample; Other: vaginal sample

INTERVENTIONS:
Other: Blood test — A blood test (2 x 5 ml dry tubes) will be taken to analyze steroid profiles
Other: urine sample — a 20 ml urine sample will be taken to analyze steroid profiles
Other: vaginal sample — to characterize the microbiota.

SUMMARY:
Endometriosis is a systemic, steroid-dependent, inflammatory disease characterized by the growth of endometrial-like tissue outside the uterus, affecting approximately 10 % of women of childbearing age. The etiology and pathophysiology of endometriosis is not completely understood to support effective treatment and prevention strategies. Despite the steroid dependency, little is known concerning the underlying metabolism of estrogen and other tightly related steroids. Moreover, shortening the long diagnostic delays is a major priority in endometriosis research.

DETAILED DESCRIPTION:
The main aim of the study will be to develop a global steroidomics analytical strategy " fit-for-purpose" to improve the knowledge of endometriosis pathophysiology and boost the identification of diagnostic biomarkers.

Therefore, in a first step, a new analytical method will be developed adapting state-of-the-art liquid chromatography coupled to high resolution mass spectrometry (LC-HRMS) approaches for steroids and its metabolites towards endometriosis research. The investigators will ensure the characterization of established steroids and its metabolites known to be relevant to endometriosis, but also expand the panel with non-targeted methods to identify phase-1 and -2 metabolites potentially informing of novel steroidogenic pathways in serum and urine.

In a second phase, a case-control study will be conducted to apply the strategy in a sample of women with and without endometriosis. In a third step, the investigators will explore statistical differences in steroid profiles among endometriosis groups and evaluate the discriminative performance.

The proposed method has large applications in endometriosis research and large potential to provide novel clues about the still poorly understood steroid metabolism disruption undergoing in endometriosis. Ultimately, non-invasive biomarker discovery in urine could revolutionize endometriosis diagnosis and management, allowing for earlier detection and personalized treatment strategies, ultimately improving the lives of individuals affected by this often overlooked but debilitating condition.

In parallel, the role of dysbiosis of the vaginal microbiota on hormonal alterations linked to endometriosis will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45
* Free, informed and written consent from the patient to participate in the study
* Good understanding of the French language
* Patient affiliated to or benefiting from a social security or similar scheme

Specific inclusion criteria for each group:

Group 1. Controls.

* Women with no laparoscopically confirmed signs suggestive of deep endometriosis.
* No clinico-biological criteria in favour of a diagnosis of endometriotic disease, nor any radiological signs (ultrasound or MRI) suggestive of endometriosis.

Group 2. Cases of deep endometriosis.

* Newly diagnosed women (less than 12 months).
* Severe, deep endometriotic pathology with surgical indication (clinical examination, imaging tests, pre-operative findings).

Exclusion Criteria:

* Intercurrent diagnosis of pregnancy.
* Presence of other hormone-dependent pathologies (e.g. breast cancer, PCOS).
* Acute infection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The STERONLINE study population will be made up of women aged between 18 years and 45 years
  * 45 patients with endometrioma
  * 45 patients without endometrioma
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Identify steroid profiles associated with endometriosis | Sampling at inclusion visit
  Statistical associations between steroids and the presence of endometriosis.

SECONDARY OUTCOMES:
Identify biomarkers of environmental chemical exposure associated with endometriosis and steroid profiles. | Sampling at inclusion visit
  Statistical difference between environmental chemical and steroid exposure profiles between subgroups of the study populations.
Identify the role of vaginal microbiota dysbiosis on hormonal alteration in endometriosis | Sampling at inclusion visit
  Presence of a specific bacterial community in the vaginal microbiota

IPD SHARING:
Plan to Share IPD: Yes